CLINICAL TRIAL: NCT05106764
Title: Early Detection of Fabry Disease (FD): Using Real-World Data for the Development of Advanced Natural Language Processing Methods: Retrospective Database Analysis
Brief Title: Early Detection of Fabry Disease
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-675-4011-1; FLAGGING FD-1 (Other: Takeda)
Record Dates: First submitted 2021-10-25; First posted 2021-11-04 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Fabry Disease
MeSH Terms: conditions — Fabry Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Retrospective Database Analysis: Data from patient's hospital records of the last 10 years will be collected/extracted retrospectively using epidemiological methods to test the forecasting power of the algorithm.
  Interventions: Other: No intervention

INTERVENTIONS:
Other: No intervention — This is non-interventional study.

SUMMARY:
The main aim of this study is early detection of FD using real-world data for the development of advanced natural language processing methods and to develop a predictive algorithm and to measure the performance of the algorithm in identifying participants with FD.

This study is about using data from hospital Electronic Health Record database from the last 10 years to describe the ranking of participants with FD using multilevel likelihood ratios and to validate the algorithm using positive controls. No investigational medicinal product or device will be tested in this study. Hospital electronic health record data will be analyzed for a period of up to 6 months.

ELIGIBILITY:
Inclusion criteria:

* In-patient or out-patient datasets of the participating hospital in the last 10 years
* Participants at any age Positive controls: a subset of all participant hospital records that includes the participants with confirmed FD.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Data from all in-patient or out- patient datasets of the participating hospital in the last 10 years will be used to test the forecasting power of the algorithm.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2023-11-30 (Actual); Primary Completion 2025-12-16 (Actual); Study Completion 2025-12-16 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Positive Predictive Value (PPV) at Different Cut-off Values (top 10, 20, 50, 100 and 200) | Up to End of the study (approximately 6 months)
  PPV is a clinically relevant statistical measure that indicates how likely participants that screen positive are to be affected by the condition assessed. Thus, the PPV can be considered as the percentage of participants which are identified as FD candidates by the ranking algorithm who are indeed FD participants. As FD predictive algorithm, we will use (multilevel) likelihood ratios (LRs) as this method permits a good use of clinical test results to establish diagnoses for the individual participant. LR is calculated, defined as the probability of a patient who has FD to present with this feature divided by the probability of a participant who not has FD to present with the feature: Likelihood ratio= features the participant/Fabry divided by features the participant/not Fabry. Positive predictive value of the algorithm at several cutoffs (top 10, top 20, top 50, top 100, top 200) will be reported.

SECONDARY OUTCOMES:
Percentage of Participants Based on Ranking With Known FD Using Multilevel Likelihood Ratios For Algorithm Validation Purposes | Up to End of the study (approximately 6 months)
  To validate the algorithm, records of participants with a high predictive value are reexamined by medical experts who assess the likelihood of FD based on the participant records. Percentage of participants based on ranking with known FD using multilevel likelihood ratios for algorithm validation purpose will be reported. Likelihood ratio= features the participant/Fabry divided by features the participant/not Fabry.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (3):
- Germany (3):
  - Universitätsklinikum Erlangen Kinder- und Jugendklinik, Erlangen
  - Universitätsklinikum Erlangen Neurologische Klinik, Erlangen
  - Universitätsmedizin Mainz Villa Metabolica Zentrum für Kinder- und Jugendmedizin, Mainz

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/61bcf691f571d4002a64b4b7